CLINICAL TRIAL: NCT04177602
Title: Evaluating Trifluridine/Tipiracil Based Chemoradiation in Locally Advanced Rectal Cancer - The Phase I/II TARC Trial
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the amended therapy strategies for rectal cancer recently, it was decided not to transfer the study to the phase II part, as superiority over standard chemoradiation and transfer to a new therapy standard are increasingly unlikely.
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Clinical Trial Center North (CTC North GmbH & Co. KG) (Other); Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TARC-01
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: trifluridine tipiracil chemoradiation; locally advanced rectal cancer; neoadjuvant; adenocarcinoma of the rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Trifluridine

STUDY DESIGN:
Intervention Model Description: Seamless phase I/II trial with phase I part for determination of maximum tolerated dose (MTD) of Trifluridine/tipiracil, followed by a randomized phase II trial (randomization ratio 2:1) with an experimental arm with Trifluridine/tipiracil based chemoradiotherapy (CRT) and a standard - calibration arm (internal control) with capecitabine CRT flanked by translational research
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trifluridine/tipiracil based radiotherapy (Experimental): Trifluridine/tipiracil based chemoradiotherapy (CRT)
  Interventions: Combination Product: Trifluridine/tipiracil chemoradiation
- standard calibration arm (internal control) (Active Comparator): capecitabine based chemoradiotherapy
  Interventions: Combination Product: Capecitabine based chemoradiation

INTERVENTIONS:
Combination Product: Trifluridine/tipiracil chemoradiation — Trifluridine/tipiracil based chemoradiation
  Arms: Trifluridine/tipiracil based radiotherapy
Combination Product: Capecitabine based chemoradiation — Capecitabine based chemoradiation
  Arms: standard calibration arm (internal control)

SUMMARY:
Seamless phase I/II trial with phase I part for determination of maximum tolerated dose (MTD) of Trifluridine/tipiracil, followed by a randomized phase II trial (randomization ratio 2:1) with an experimental arm with Trifluridine/tipiracil based chemoradiotherapy (CRT) and a standard - calibration arm (internal control) with capecitabine CRT flanked by translational research in patients with locally advanced rectal cancer

DETAILED DESCRIPTION:
This is a multicenter randomized seamless phase I/II trial with a phase I for determination of maximum tolerated dose (MTD) of Trifluridine/tipiracil, followed by a randomized phase II trial (randomization ratio 2:1) with an experimental arm with Trifluridine/tipiracil in combination with standard radiotherapy and a standard - calibration arm (internal control) with capecitabine CRT flanked by translational research, designed to assess the clinical performance and efficacy of Trifluridine/tipiracil compared to current standard capecitabine chemoradiation in patients with locally advanced rectal cancer.

The primary clinical objective in phase I is to determine the dosage and feasibility of Trifluridine/tipiracil based chemoradiation and in phase II whether Trifluridine/tipiracil with preoperative chemoradiation improves pathological complete remissions in patients with locally advanced rectal cancer.

The secondary objectives are to evaluate Trifluridine/tipiracil chemoradiation with respect to disease free survival, overall survival, local regional failure, pathological down-staging (ypT0-2N0) rate, tumour regression grade, histopathological R0 resection rate, neoadjuvant rectal score (NAR), and perioperative complication rate. Safety and toxicity, according to NCI CTC AE v5, quality of life and feasibility of the regimen are further secondary objectives that are to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with histologically proven adenocarcinoma of the rectum (tumour ≤ 12 cm from the anal verge)
2. Indication for neoadjuvant chemoradiation: clinical tumour stage T3/4 or any node-positive disease (clinical stage according the TNM classification system, based on MRI).
3. No evidence of metastatic disease (as evidenced by negative CT-scan of the chest and abdomen).
4. The disease must be considered either resectable at the time of entry or expected to become resectable after preoperative chemoradiation.
5. Age ≥ 18 years
6. WHO/ECOG Performance Status ≤ 2
7. No prior cytotoxic chemotherapy or radiotherapy for rectal cancer.
8. No prior radiotherapy to the pelvis, for any reason.
9. Presence of adequate contraception in fertile patients. Adequate methods of contraception are: intra-uterine device, hormonal contraception, condom use with spermicide. Pregnant or breastfeeding women are excluded from participation.
10. Adequate bone marrow, hepatic and renal function: Haemoglobin ≥9.0 g/dL (transfusions allowed to achieve or maintain levels), absolute neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, ALAT, ASAT ≤ 2.5 x ULN, Alkaline phosphatase ≤ 2.5 x ULN, Total bilirubin ≤1.5 x ULN, Creatinine clearance > 50 mL/min (calculated according to Cockroft and Gault).
11. Ability to swallow tablets.
12. Written informed consent and patient's agreement to comply with the study protocol.

Exclusion Criteria:

1. Previous (within the last 3 years) or concurrent malignancies, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix or basal cell carcinoma of the skin.
2. Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia not well controlled with medication) or myocardial infarction within the last 12 months.
3. Known allergy or any other adverse reaction to any of the study drugs or to any related compound.
4. Known significant impairment of intestinal resorption (e.g. chronic diarrhea, inflammatory bowel disease).
5. Pre-existing condition which would deter chemoradiotherapy or radiotherapy, i.e. fistulas, severe ulcerative colitis (particularly patients currently taking sulphasalazine), Crohn's disease, prior adhesions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD)/Phase 1 part | 8 weeks
  Toxicity
Rate of pathological complete remissions (pCR)/Phase 2 part | 3 months
  Pathohistological response

SECONDARY OUTCOMES:
Disease free survival (DFS) | 4 years
  recurrence and survival
Overall survival (OS) | 4 years
  Survival
Loco-regional failure | 4 years
  Loco-regional recurrence
Histopathological R0 resection rate | 3 months
  Pathohistological response
Tumour regression grades | 3 months
  Pathohistological response
Pathological down-staging (ypT0-2N0) rate | 3 months
  Pathohistological response
Neoadjuvant rectal score (NAR) | 3 months
  Clinical stage and Pathohistological response (<8 low, 8-16 intermediate, >16 high risk)
Adverse event rate | 3 months
  Rate of adverse events according to NCI CTC AE v5
Rate of perioperative complications | 3 months
  Perioperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stein, Principal Investigator — University Cancer Center Hamburg
Locations (8):
- Germany (8):
  - Malteser Krankenhaus St. Franziskus Hospital, Flensburg, Schleswig-Holstein
  - Lübecker Onkologische Schwerpunktpraxis Dres. med. Uthgenannt, Kirso, Weber, Lübeck, Schleswig-Holstein
  - Klinik Dr. Hancken / MVZ Onkologie, Stade, Schleswig-Holstein
  - University Medical Center Halle, Halle
  - Hämatologisch- Onkologische Praxis Eppendorf (HOPE), Hamburg
  - II. Medizinische Klinik und Poliklinik Hubertus Wald Tumorzentrum - UCCH, Hamburg
  - Überörtliche Gemeinschaftspraxis für Innere Medizin Schwerpunkt Hämatologie, Onkologie und Palliativmedizin Dres. Verpoort, Wierecky & Zeller, Hamburg
  - Hämatologisch- Onkologische Praxis Altona (HOPA), Hamburg

REFERENCES:
- [Derived] Thiele B, Stein A, Schultheiss C, Paschold L, Jonas H, Goekkurt E, Russel J, Schuch G, Wierecky J, Sinn M, Tintelnot J, Petersen C, Rothkamm K, Vettorazzi E, Binder M. Trifluridine/Tipiracil Based Chemoradiation in locally Advanced Rectal Cancer: The Phase I/II TARC Trial. Clin Colorectal Cancer. 2025 Mar;24(1):11-17. doi: 10.1016/j.clcc.2024.06.003. Epub 2024 Jun 22. PMID 39003182
- [Derived] Rothkamm K, Christiansen S, Rieckmann T, Horn M, Frenzel T, Brinker A, Schumacher U, Stein A, Petersen C, Burdak-Rothkamm S. Radiosensitisation and enhanced tumour growth delay of colorectal cancer cells by sustained treatment with trifluridine/tipiracil and X-rays. Cancer Lett. 2020 Nov 28;493:179-188. doi: 10.1016/j.canlet.2020.08.038. Epub 2020 Sep 4. PMID 32891715